CLINICAL TRIAL: NCT04478838
Title: "Re-examining Maintenance Antipsychotic Treatment in Schizophrenia: "Extended" Antipsychotic Dosing"
Brief Title: "Extended" (Alternate Day) Antipsychotic Dosing
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Gary Remington, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 154-2018
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2024-07

CONDITIONS: Schizophrenia and Related Disorders; Drug Administration Schedule; Drug Therapy; Antipsychotic Agents
Keywords: Extended Dosing; Alternate day dosing; Olanzapine; Risperidone; Paliperidone
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Olanzapine; Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended Dosing Group (Experimental): Participants taking olanzapine or risperidone or paliperidone will be switched to an alternate day dosing schedule.
  Interventions: Drug: Risperidone; Drug: Olanzapine; Drug: paliperidone
- Treatment as Usual group (No Intervention): Participants will continue to take their olanzapine or risperidone or paliperidone following the same prescribed daily schedule.

INTERVENTIONS:
Drug: Risperidone — 0.25 mg, 0.5 mg, 1 mg, 2 mg, 3 mg and 4 mg Tablets
  Other Names: Risperdal
  Arms: Extended Dosing Group
Drug: Olanzapine — 2.5 mg, 5 mg, 7.5 mg, 10 mg, 15 mg, 20 mg Tablets
  Other Names: Zyprexa; Apo-Olanzapine; Sandoz-Olanzapine
  Arms: Extended Dosing Group
Drug: paliperidone — 3 mg, 6 mg, 9 mg Tablets
  Other Names: Invega
  Arms: Extended Dosing Group

SUMMARY:
The study wishes to examine whether "extended" antipsychotic treatment, in this case, antipsychotic treatment every other day, is as effective as daily treatment. It is also evaluating whether there may be differences in terms of side effects.

Participants will be randomly assigned to either the treatment as usual group (i.e., taking antipsychotic daily) or the extended dosing group (i.e., taking antipsychotic one day on, one day off). That means, like flipping a coin, there is a 50/50 chance that participants will continue on daily dosing of your antipsychotic or have it switched to every other day dosing.

This study will last for 1 year. Participants will be evaluated at the beginning and every two weeks during the first 6 months, with visits once every 4 weeks for the final 6 months. In total, participants will make 22 visits over 52 weeks to the investigator's office.

The investigators hypothesize that with ED, there will be no change in symptom severity but improvement in the frequency and severity of side effects, wellbeing, and functioning.

DETAILED DESCRIPTION:
This is a randomized, double-blind, controlled trial that will compare ED, i.e. alternate day dosing to daily dosing i.e. TAU.

Individuals will be randomized to ED or TAU using a permuted block design with a random number generator. The size will be fixed and study personnel blinded to the randomization block size.

To maintain a double-blind design, our pharmacy will provide, on an individualized basis, APs at the appropriate dose and placebo where necessary in matching gelatin capsules, packaged in blister packs. The active tablet will be over-encapsulated, and matching placebo will be prepared using the same capsules (filled with lactose). Thus, from the individual subject's position, AP treatment is continued according to the same daily schedule. Further, if their current medication is prescribed in divided doses, this too will be employed during the study. The minimum and maximum doses for Risperidone will be 1 mg and 16mg respectively. The minimum and maximum doses for Olanzapine will be 5 mg and 20mg respectively. The minimum and maximum doses for Paliperidone will be 3 mg and 12mg respectively. Other psychotropic medications prescribed before the study will be permitted, with any changes in dosing during its course documented

The trial is 1 year in duration. To prevent bias, the study code will remain blinded until the trial's completion.

Study visits will be scheduled every 2 weeks over the first 6 months, in line with the earlier investigation. Thereafter, the visits will be decreased to every 4 weeks, aligning with the schedule routinely observed in our ambulatory clinics.

The investigators are asking the following questions:

1. (Non-inferiority) Can additional confirmatory evidence support "extended" AP dosing (ED) as an alternative to continuous administration, i.e. is it as effective clinically?
2. (Superiority) Can the investigators establish clinical benefits (e.g. better tolerability, fewer side effects, such as decreased glucose dysregulation) with ED?

Hypothesis: The investigators hypothesize that with ED, there will be no change in symptom severity but improvement in the frequency and severity of side effects, wellbeing, and functioning.

ELIGIBILITY:
Inclusion Criteria:

(i) A primary diagnosis of a Schizophrenia Spectrum or Other Psychotic Disorder as defined by the DSM-5 diagnosis and confirmed by the MINI (Version 7.0.2)

(ii) age 18 or older

(iii) female participants of childbearing potential must be using a reliable method of contraception and have a negative pregnancy test at the time of enrolment and must, in the investigator's opinion, practice a clinically accepted, reliable method of contraception during this study. Male participants must not father a baby during their time in the study

(iv) ability to communicate in English

(v) capacity to provide written, informed consent, as assessed using the MacCAT-CR at time of consent

(vi) stabilized as outpatients with a single oral AP (risperidone or olanzapine or paliperidone*) at the same dose for ≥3 months i. On a prescribed risperidone dose of between 1-6mg, or a prescribed olanzapine dose of between 5-20mg, or a prescribed paliperidone 3-12mg

(vii) evidence of adherence with current AP treatment

Exclusion Criteria:

(i) exposure to a depot AP within 1 year (i.e., no depot AP injection within the last year)

(ii) Current diagnosis of substance use disorder according to DSM-5 criteria (verified through the MINI for Psychotic Disorders (Version 7.0.2) and a positive drug screen for street and /or prescription drugs not prescribed to the participant by treating physicians

(iii) ECT within the last 3 months

(iv) pregnancy or lactation

(v) neurological condition (dementia including Alzheimer's disease, multiple sclerosis, epilepsy, stroke, or traumatic brain injury)

(vi) allergy to the study drugs and their excipients

(vii) allergy (e.g., galactosaemia) or severe intolerance to lactose

(viii) negative urine drug screen result for Olanzapine or Risperidone or Paliperidone (if applicable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Deterioration using the "Brief Psychiatric Rating Scale - Expanded" | 0 and 52 weeks
  Change in the Brief Psychiatric Rating Scale - total scores from baseline to 52 weeks. The score values for each item on the BPRS range from 1 to 7. The higher the score for each item the worse the outcome. The values for each item on the BPRS are scored as follows:
  1- Not Present, 2 - Very Mild, 3- Mild, 4- Moderate, 5 - Moderately Severe, 6- Severe, 7- Very Severe.

SECONDARY OUTCOMES:
Exploratory Outcomes - Symptoms 1 using "The Clinical Global Impression - Schizophrenia Scale" | 0 and 52 weeks
  Change in Clinical Global Impression - Schizophrenia (CGI-SCH) severity of illness scores from baseline to 52 weeks. The severity of illness score values for each item on the CGI- SCH range from 1 to 7. The higher the score for each item the worse the outcome.
  The severity of illness values are scored as follows:
  1- Normal, not ill, 2 -Minimally ill, 3- Mildly ill, 4- Moderately ill, 5 - Markedly ill, 6- Severely ill, 7- Among the most severely ill.
Exploratory Outcomes - Symptoms/Side Effects using "The Clinical Global Impression - Schizophrenia Scale" | 0 and 52 weeks
  Change in Clinical Global Impression - Schizophrenia Scale (CGI-SCH) degree of change scores from baseline to 52. The values range from 1-7. The higher the score for each item the worse the outcome. The score value of each item are as follows:
  1 - Very much improved, 2 - Much Improved, 3 - Minimally improved, 4 - No Change, 5 - Minimally Worse, 6- Much Worse, 7 - Very Much Worse
Exploratory Outcomes - Symptoms 3 using the "Calgary Depression Scale for Schizophrenia" | 0 and 52 weeks
  Change in Calgary Depression Scale (CDS) scores from baseline to 52 weeks. Scores range from 0-3 as follows: 0- Absent, 1- Mild, 2- Moderate, 3 - Severe. The higher the score for each item, the worse the outcome.
Exploratory Outcomes - Symptoms 4 using the "Yale-Brown Obsessive-Compulsive Scale" | 0 and 52 weeks
  Change in Yale-Brown Obsessive-Compulsive Scale (YBOCS) scores from baseline to 52 weeks. Scores range from 0-4 with higher scores indicating worsening of outcome.
Exploratory Outcomes - Symptoms 5 using the "Hamilton Anxiety Scale" | 0 and 52 weeks
  Change in Hamilton Anxiety Scale (HAM-A) scores from baseline to 52 weeks. Scores on each item range from 0-4 as follows: 0- not present, 1- mild, 2 - moderate, 3- severe, 4 - very severe. Higher scores on each item and total score indicate worsening of anxiety outcome.
Exploratory Outcomes - Side Effects 1 using the "Leibowitz Social Anxiety Scale" | 0 and 52 weeks
  Change in Liebowitz Social Anxiety Scale (LSAS) scores from baseline to 52 weeks. For each item, there are 2 scores; 1) score for fear of anxiety and 2) score for avoidance. For the fear of anxiety component of the scale, score ranges from 0-3 as follows: 0- None, 1- Mild, 2- Moderate, 3 - Severe. The scores for the Avoidance component of the scale ranges from 0-3 as follows: 0 - Never, 1- Occasionally, 2 - Often, 3 - Usually. The higher the score the worse the outcome.
Exploratory Outcomes - Side Effects 2 using the "Neurological Evaluation Scale" | 0 and 52 weeks
  Change in Neurological Evaluation Scale (NES) scores from baseline to 52 weeks. There are 12 items and scores for each item range from 0-2 with higher scores indicating worsening of outcome. Item 5 does not require a score.
Exploratory Outcomes - Side Effects 3 using the "Glasgow Assessment Side-Effect Scale" | 0 and 52 weeks
  Change in Glasgow Assessment Side-Effect Scale (GASS) scores from baseline to 52 weeks. Scores range from 0-3 as follows: 0 -Never, 1- Once, 2 - A few times, 3 - Everyday. The higher the score for each item and higher total indicates a worse side effect outcome.
Exploratory Outcomes - Side Effects 4 using the "Drug Attitude Inventory" Scale | 0 and 52 weeks
  Change in Drug Attitude Inventory (DAI) scores from baseline to 52 weeks. Scores are based on 30 true/false statements.There are 15 items that a patient who is fully adherent to their prescribed medication (and so would be expected to have a positive response to medication would answer true and 15 items such a patient would answer as false. Each positive answer is given a score of plus one, and each negative answer is given a score of minus one. The total positive score would indicate a positive response (adherent to medication) whereas a negative total score would indicate a negative response (non adherent to medication).
Exploratory Outcomes - Side Effects 5 using the "Barnes Akathisia Rating Scale" | 0 and 52 weeks
  Change in Barnes Akathisia Rating Scale (BARS) scores from baseline to 52 weeks. The total score for the global clinical assessment of akathisia ranges from 0-5 with higher score indicating a worsening of akathisia.
Exploratory Outcomes - Side Effects 6 using the "Simpson Angus Scale" | 0 and 52 weeks
  Change in Simpson Angus Scale (SAS) scores from baseline to 52 weeks. There are 13 items in the scale; scores on each item range from 0-4 with higher scores indicating worse extrapyramidal outcome.
Exploratory Outcomes - Side Effects 7 using the "Abnormal Involuntary Movement Scale" | 0 and 52 weeks
  Change in Abnormal Involuntary Movement Scale (AIMS) scores from baseline to 52 weeks. There are 13 items in the scale, scores on each item range from 0-4 with higher scores indicating a worse outcome in abnormal movements.
Exploratory Outcomes - Wellbeing using the "Quality of Life and Satisfaction Questionnaire" | 0 and 52 weeks
  Change in Quality of Life Scale (QLS) scores from baseline to 52 weeks. The scores for each item range from 0-6. The higher the score, the better the outcome. On several items, there is an additional score of "9" to indicate "not applicable".
Exploratory Outcomes - Wellbeing 2 using the "Quality of Life and Satisfaction Questionnaire - Short Form" | 0 and 52 weeks
  Change in Quality of Life and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) scores from baseline to 52 weeks. Scores range from 0-6 with lower scores indicating a worse outcome.
Exploratory Outcomes - Wellbeing 3 using the "Subject Happiness Scale" | 0 and 52 weeks
  .Change in Subjective Happiness Scale (SHS) scores from baseline to 52 weeks. There are 4 items; scores on each item range from 1-7 with higher scores indicating a happier outcome.
Exploratory Outcomes - Function 1 using the "Social and Occupational Function Assessment Scale" | 0 and 52 weeks
  Change in : Social and Occupational Function Assessment Scale (SOFAS). scores from baseline to 52 weeks. A total score ranges from 0-100 with higher scores indicating better social and occupational functioning..
Exploratory Outcomes - Function 2 using the "Personal and Social Performance Scale" | 0 and 52 weeks
  Change in Personal and Social Performance scale (PSP) scores from baseline to 52 weeks. The ratings are based on four areas (a) socially useful activities, including work and study; b) personal and social relationships; c) self, and d) disturbing and aggressive behaviours. Overall score range from 1-100. The higher the overall rating, the better the outcome. The breakdown of the total Rating score are as follows: scores ranging from 1-30 reflect functioning so poor that intensive support or supervision is needed; ratings from 31-70 reflect manifest disabilities of various degrees; ratings from 71-100 reflect only mild difficulties.
Exploratory Outcomes - Function 3 using the "Recovery Assessment Scale" | 0 and 52 weeks
  Change in Recovery Assessment Scale (RAS) scores from baseline to 52 weeks. There are 41 items with scores on each item ranging from 1-5 with higher scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Gary J Remington, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No